CLINICAL TRIAL: NCT01472913
Title: Fibrin Sealant in Bilateral Simultaneous Total Knee Arthroplasty. A Prospective Randomised Double-blinded Study Focus in on: Blood Loss, Pain, ROM, Swelling and Strength
Brief Title: Fibrin Sealant in Bilateral Simultaneous Total Knee Arthroplasty With Focus on Blood Loss, Pain, Swelling and Strength
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Christian Skovgaard Nielsen, M.D. Orthopedic Surgery, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-A-2009-69
Record Dates: First submitted 2011-10-11; First posted 2011-11-17 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Blood Loss
Keywords: Prospective randomised double-blind study; Fibrin sealant; Bilateral simultaneous total knee arthroplasty; Blood loss; Postoperative pain; Complications
MeSH Terms: conditions — Hemorrhage; Pain, Postoperative | interventions — Fibrin Tissue Adhesive; Saline Waters

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fibrin Sealent (Active Comparator)
  Interventions: Drug: Fibrin sealant
- Saline water (Placebo Comparator)
  Interventions: Drug: Saline water

INTERVENTIONS:
Drug: Fibrin sealant — Fibrin sealant is applied on the surfaces of bone and soft tissue of surgery after placement of the prothesis due to the randomised knee.
  Other Names: Evicel, ATC-kode B02BC30
  Arms: Fibrin Sealent
Drug: Saline water — Same procedure to the opposite knee (the same patient) performed with sprayed saline water (placebo).
  Arms: Saline water

SUMMARY:
The purpose of this study is to measure the effect of fibrin sealant on reducing blood loss, pain and swelling when operated for bilateral total knee arthroplasty. Likewise the effect on Range Of Movement (ROM) and strength is examined.

ELIGIBILITY:
Inclusion Criteria:

* Elective bilateral knee arthroplasty
* Must speak and understand Danish
* Musk be able to gave oral and written consent.
* Females must be post-menopausal, and last menstruation must be minimum of one year ago.

Exclusion Criteria:

* Alcohol or medicine abuse
* Treatment with opioids
* Allergy to local anaesthetics
* Allergy to active substances i fibrin sealant
* Age below 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-08; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Blood loss | 24 hours postoperative
  24 hours postopertive blood loss estimated by drains from each of the knees .

SECONDARY OUTCOMES:
Pain | 2-3 weeks before the operation and on 1st, 2nd, 3rd, 7th and 21st postoperative day.
  2-3 weeks before surgery the patients participate in an information meeting likewise the patients are tested for all secundary outcomes by a physiotherapist.
  Measurement of postoperative pain is done on the 1st, 2nd and 3rd day before mobilization. On the 7th and 21st postoperative day the majority of the patients are discharged and therefore testet at the outpatient department.
swelling | 2-3 weeks before surgery and 1st, 2nd, 3rd, 7th and 21st postoperative day
  2-3 weeks before surgery the patients participate in an information meeting likewise the patients are tested for all secundary outcomes by a physiotherapist.
  Measurement of postoperative swelling is done on the 1st, 2nd and 3rd day before mobilization. On the 7th and 21st postoperative day the majority of the patients are discharged and therefore testet at the outpatient department. The swelling is measured as the difference of circumference 1 cm proximal of the patella 2-3 weeks before surgery and at the outlined postoperative times.
Range of Movement (ROM) | 2-3 weeks before surgery and on the 3rd, 7th and 21st postoperative day
  2-3 weeks before surgery the patients participate in an information meeting likewise the patients are tested for all secondary outcomes by a physiotherapist.
  Measurement of postoperative ROM is done on the 3rd day before mobilization. On the 7th and 21st postoperative day the majority of the patients are discharged and therefore testet at the outpatient department.
Strength | 2-3 weeks before the operation and on the 3rd, 7th and 21st postoperative day
  2-3 weeks before surgery the patients participate in an information meeting likewise the patients are tested for all secondary outcomes by a physiotherapist.
  Measurement of postoperative strength is done on the 3rd day before mobilization. On the 7th and 21st postoperative day the majority of the patients are discharged and therefore testet at the outpatient department.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Skovgaard Nielsen, M.D, Principal Investigator — Hvidovre University Hospital; Henrik Husted, M.D., Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark